CLINICAL TRIAL: NCT05421572
Title: Epidemiological Survey on Metabolic Dysfunction-Associated Fatty Liver Disease (MAFLD)
Acronym: MAFLD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Tsinghua Chang Gung Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CG-MAFLD-001
Record Dates: First submitted 2022-06-06; First posted 2022-06-16 (Actual); Last update posted 2022-06-16 (Actual); Status verified 2022-05

CONDITIONS: Fatty Liver Disease
Keywords: MAFLD
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single Group Assignment: Adults with health check-ups at multiple health examination centers across China
  Interventions: Diagnostic Test: Fibrotouch

INTERVENTIONS:
Diagnostic Test: Fibrotouch — Fibrotouch will be performed showing the stiffness and fat content of liver

SUMMARY:
To investigate the prevalence of Metabolic Dysfunction-Associated Fatty Liver Disease (MAFLD) among adults in China

DETAILED DESCRIPTION:
Non-Alcoholic Fatty Liver Disease (NAFLD) is the most common chronic liver disease all over the world (1). In early 2020, a new definition of MAFLD has been proposed and is becoming increasingly widely accepted. The new diagnostic criteria are based on the histology or imaging of liver biopsies, or even blood biomarker tests indicative of the presence of fatty liver while satisfying any one of the following three conditions: overweight/obesity, type 2 diabetes, or metabolic dysfunction (2). The information on the prevalence of MAFLD is scarce. This study is designed to conduct MAFLD screening in adults with health check-ups at multiple health examination centers across China. The primary objective is to investigate the prevalence of MAFLD among adults in China.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 75, both sex;
* Able to sign informed consent.

Exclusion Criteria:

* Pregnant women and those who are implanted with pacemakers, stents or any other metal devices.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: adults with health check-ups at multiple health examination centers across China.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2022-06-10 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
To investigate the prevalence of MAFLD among adults at multiple health examination centers across China. | through study completion, an average of 1 year
  MAFLD means metabolic dysfunction-associated fatty liver disease

SECONDARY OUTCOMES:
To assess the proportion of overweight or obese patients with MAFLD (BMI≥23 kg/m²). | through study completion, an average of 1 year
  MAFLD means metabolic dysfunction-associated fatty liver disease; BMI means body mass index
To assess the prevalence of metabolic dysfunction among patients with MAFLD who are lean or normal in body weight (BMI < 23 kg/m²) | through study completion, an average of 1 year
  MAFLD means metabolic dysfunction-associated fatty liver disease; BMI means body mass index
To assess the prevalence of type 2 diabetes among patients with MAFLD. | through study completion, an average of 1 year
  MAFLD means metabolic dysfunction-associated fatty liver disease
To assess the prevalence of liver fibrosis and cirrhosis among patients with MAFLD. | through study completion, an average of 1 year
  MAFLD means metabolic dysfunction-associated fatty liver disease

CONTACTS AND LOCATIONS:
Locations (1):
- Bejing Tsinghua Chang Gung Hospital, Beijing, Bejing, China

IPD SHARING:
Plan to Share IPD: Undecided
Not yet determined

REFERENCES:
- [Background] Younossi ZM, Koenig AB, Abdelatif D, Fazel Y, Henry L, Wymer M. Global epidemiology of nonalcoholic fatty liver disease-Meta-analytic assessment of prevalence, incidence, and outcomes. Hepatology. 2016 Jul;64(1):73-84. doi: 10.1002/hep.28431. Epub 2016 Feb 22. PMID 26707365
- [Background] Eslam M, Newsome PN, Sarin SK, Anstee QM, Targher G, Romero-Gomez M, Zelber-Sagi S, Wai-Sun Wong V, Dufour JF, Schattenberg JM, Kawaguchi T, Arrese M, Valenti L, Shiha G, Tiribelli C, Yki-Jarvinen H, Fan JG, Gronbaek H, Yilmaz Y, Cortez-Pinto H, Oliveira CP, Bedossa P, Adams LA, Zheng MH, Fouad Y, Chan WK, Mendez-Sanchez N, Ahn SH, Castera L, Bugianesi E, Ratziu V, George J. A new definition for metabolic dysfunction-associated fatty liver disease: An international expert consensus statement. J Hepatol. 2020 Jul;73(1):202-209. doi: 10.1016/j.jhep.2020.03.039. Epub 2020 Apr 8. PMID 32278004